CLINICAL TRIAL: NCT03597529
Title: CHOCOlate MeLatonin for AdolescenT MigrainE: The CHOCOLATE Study
Brief Title: CHOCOlate MeLatonin for AdolescenT MigrainE
Acronym: CHOCOLATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amy Gelfand (Other)
Responsible Party: Sponsor-Investigator, Amy Gelfand, Assistant Professor of Neurology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-22645
Record Dates: First submitted 2017-06-26; First posted 2018-07-24 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-Dose Melatonin (mg) (Experimental): melatonin 2mg (equal to or over 40kg) melatonin 1mg (under 40kg) Melatonin: melatonin
  Interventions: Drug: Melatonin
- High-Dose Melatonin (mg) (Experimental): melatonin 8mg (equal to or over 40kg) melatonin 4mg (under 40kg) Melatonin: melatonin
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — melatonin

SUMMARY:
Existing treatments for acute migraine are not effective for all children and adolescents, and can cause side effects. Investigator propose a dose-finding study of melatonin for acute migraine treatment in children and adolescents to determine the best dose to bring forward in a future fully-powered efficacy trial.

DETAILED DESCRIPTION:
This pilot randomized trial is a dose-finding study to determine which dose of melatonin is most effective for treating acute migraine in children and adolescents who have episodic migraine. Investigator will identify the most effective dose to pull forward into a future fully-powered placebo-controlled efficacy study. If both doses are equally effective, Investigator will bring forward the best tolerated dose. If doses are equally well tolerated, Investigator will bring forward the lowest effective dose, as this will minimize cost to families should this treatment become widely adopted.

ELIGIBILITY:
Inclusion Criteria:

1. Meet ICHD criteria for episodic migraine in children and adolescents, with at least 1 migraine attack per month on average.
2. Age 3-17 years
3. Dissatisfaction with previous acute treatments, for one or more of the following reasons: a) One or more previously tried acute medications have not been effective, or adequately effective, b) previously tried acute treatments have caused side effects, or C) patient/family would prefer a natural supplement for acute treatment over medication treatment
4. If of driving age, teen participant agrees not to drive for at least 8 hours after treating with melatonin.

Exclusion Criteria:

1. Allergy or intolerance to melatonin, or to chocolate.
2. Opioid or barbiturate overuse as defined in ICHD
3. Pregnant/lactating

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Gelfand, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Victor TW, Hu X, Campbell JC, Buse DC, Lipton RB. Migraine prevalence by age and sex in the United States: a life-span study. Cephalalgia. 2010 Sep;30(9):1065-72. doi: 10.1177/0333102409355601. Epub 2010 Mar 12. PMID 20713557
- [Background] Ambriz-Tututi M, Rocha-Gonzalez HI, Cruz SL, Granados-Soto V. Melatonin: a hormone that modulates pain. Life Sci. 2009 Apr 10;84(15-16):489-98. doi: 10.1016/j.lfs.2009.01.024. Epub 2009 Feb 15. PMID 19223003
- [Background] Gitto E, Aversa S, Salpietro CD, Barberi I, Arrigo T, Trimarchi G, Reiter RJ, Pellegrino S. Pain in neonatal intensive care: role of melatonin as an analgesic antioxidant. J Pineal Res. 2012 Apr;52(3):291-5. doi: 10.1111/j.1600-079X.2011.00941.x. Epub 2011 Dec 5. PMID 22141591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ran from September 25, 2017 until November 5, 2019. Eligibility was assessed by a pediatric headache specialist.
Pre-assignment Details: Out of 102 participants who were assessed for eligibility, 84 met inclusion criteria and were randomized to a treatment.
Period: Overall Study
Arm/Group | Low-Dose Melatonin (mg) | High-Dose Melatonin (mg)
Started | 42 | 42
Follow-up | 22 | 24
Completed | 22 | 24
Not Completed | 20 | 18
Not completed — Lost to Follow-up | 10 | 12
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Non-compliant with study activities | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose Melatonin (mg) | High-Dose Melatonin (mg) | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 42 | 84
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (3.5) | 11.7 (3.6) | 11.8 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data on this baseline measurement is missing for one participant. While there are 84 participants total in the study, there is sex data for 83 participants total.
  Participants
    number analyzed (Participants) | 42 | 41 | 83
    Female | 23 | 23 | 46
    Male | 19 | 18 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84
Weight (kg) [Mean (Standard Deviation); unit: kg] | 45.7 (18.0) | 53.1 (25.6) | 49.3 (22.1)
Headache days per month (self report) [Mean (Standard Deviation); unit: days per month] | 5.5 (4.1) | 5.8 (3.4) | 5.6 (3.8)
Aura [Count of Participants; unit: Participants] — Population: Analysis population differs from the Overall number of baseline participants because data was not provided for this measure by all participants.
  Participants
    number analyzed (Participants) | 35 | 33 | 68
    (all) | 10 | 6 | 16
Reason(s) for dissatisfaction with previous acute medications [Number; unit: participants] — Some participants selected one or more reasons for dissatisfaction with previous acute medications.
  participants
    Ineffective | 9 | 8 | 17
    Side effects | 1 | 1 | 2
    Prefer natural options | 24 | 24 | 48
    Other | 14 | 9 | 23
Currently on migraine preventive [Count of Participants; unit: Participants] — Population: Analysis population differs from the Overall number of baseline participants because data was not provided for this measure by all participants.
  Participants
    number analyzed (Participants) | 38 | 35 | 73
    (all) | 19 | 14 | 33
Melatonin Dose/Weight [Mean (Standard Deviation); unit: mg/kg] | 0.04 (0.01) | 0.13 (0.03) | 0.08 (0.05)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Visual Analog Scale (VAS) Score
Description: Visual Analog Scale (VAS) score ranges from 0-10, measured in cm, 0 indicating no pain and 10 indicating the worst pain.
Time Frame: Baseline (Time 0) and 2 hours
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Low-Dose Melatonin (mg) | High-Dose Melatonin (mg)
Number analyzed (Participants) | 22 | 24
cm | -2.3 (2.1) | -2.7 (2.1)

ADVERSE EVENTS:
Time Frame: Participants were asked to report adverse events at 2 hours and at 24 hours after taking study treatment.
Description: Not all participants reported on the presence or absence of adverse events and some had more than 1 adverse event.
Arm/Group | Low-Dose Melatonin (mg) | High-Dose Melatonin (mg)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 13/19 | 17/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-Dose Melatonin (mg) (N=19) | High-Dose Melatonin (mg) (N=21)
Proportion who napped within 2 hours after treating (Nervous system disorders) | 9 | 14
Fatigue (Nervous system disorders) | 2 | 4
Weakness (Nervous system disorders) | 0 | 1
Clumsiness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT03597529/Prot_SAP_000.pdf